CLINICAL TRIAL: NCT01901965
Title: Could Contralateral Quadriceps Strength Training Attenuate the Strength Loss in the ACL-operated Knee?
Brief Title: Contralateral Strength-training After Anterior Cruciate Ligament (ACL) Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Contralateral_01
Record Dates: First submitted 2013-05-29; First posted 2013-07-17 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Muscle Weakness After Anterior Cruciate Ligament Reconstruction

ARMS (3):
- NMES (Experimental): neuromuscular electrical stimulation (NMES) of the quadriceps muscle with Kneehab
  Interventions: Behavioral: Neuromuscular electrical stimulation
- eccentric training (Experimental): unilateral eccentric resistance exercises
  Interventions: Behavioral: eccentric training
- sham NMES (Sham Comparator): neuromuscular electrical stimulation of the quadriceps muscle with intensity which causes no visible contraction or displacement of the leg (activation below motor threshold)
  Interventions: Behavioral: Neuromuscular electrical stimulation

INTERVENTIONS:
Behavioral: Neuromuscular electrical stimulation
  Arms: NMES; sham NMES
Behavioral: eccentric training
  Arms: eccentric training

SUMMARY:
The main aims of the study are (1) to examine the impact of contralateral strength training on the quadriceps muscle function after ACL surgery and (2) to compare the magnitude of cross-education induced by NMES versus eccentric strength training.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for ACL reconstruction surgery

Exclusion Criteria:

* Concomitant lower limb injury or disorder
* previous lower extremity open surgery on the contralateral lower limb
* cardiac disease
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in bilateral quadriceps muscle strength [Nm] | 1-2weeks preoperative/ 2weeks/ 8weeks/ 6month
Change in quadriceps muscle activation | 1-2 weeks preoperative/ 2weeks/ 8weeks/ 6month

SECONDARY OUTCOMES:
Change in muscle architecture | 1-2 weeks preoperative/ 2weeks/ 8weeks/ 6month
Change in self-reported questionnaire outcomes (KOOS, WOMAClk) | 1-2weeks preoperative/ 2weeks/ 8weeks/ 6 month
functional test outcomes | 6month postop
  Assessment of present functional status by means of hop tests

CONTACTS AND LOCATIONS:
Overall Officials: Nicola A Maffiuletti, PhD, Principal Investigator — Schulthess Klinik
Locations (1):
- Neuromuscular Research Laboratory, Schulthess Klinik, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Feil S, Newell J, Minogue C, Paessler HH. The effectiveness of supplementing a standard rehabilitation program with superimposed neuromuscular electrical stimulation after anterior cruciate ligament reconstruction: a prospective, randomized, single-blind study. Am J Sports Med. 2011 Jun;39(6):1238-47. doi: 10.1177/0363546510396180. Epub 2011 Feb 22. PMID 21343386
- [Background] Hortobagyi T, Scott K, Lambert J, Hamilton G, Tracy J. Cross-education of muscle strength is greater with stimulated than voluntary contractions. Motor Control. 1999 Apr;3(2):205-19. doi: 10.1123/mcj.3.2.205. PMID 10198150